CLINICAL TRIAL: NCT05632679
Title: Effects of a Personalized Sound Intervention on Anxiety, Pain, and Satisfaction During Autogenous Gingival Graft in Adults: A Randomized Controlled Trial
Brief Title: Effect of a Personalized Sound Intervention During Autogenous Gingival Grafts in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Robert Durand, Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-1146
Record Dates: First submitted 2022-09-05; First posted 2022-11-30 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Music Intervention; Gingival Graft; Anxiety; Pain; Dissatisfaction
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Single-blind randomized clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- personalized music intervention (Experimental)
  Interventions: Other: personalized music intervention
- selected audio book (Active Comparator)
  Interventions: Other: selected audio book
- standard care (No Intervention)

INTERVENTIONS:
Other: personalized music intervention — participants who are randomly selected to this group will choose three set of music they prefer among the available selection of instrumental music in the application
  Arms: personalized music intervention
Other: selected audio book — participants who are randomly selected to this group will choose one audio book they prefer among the available selection of audio books on the tablet
  Arms: selected audio book

SUMMARY:
Anxiety feeds the avoidance of dental treatments, leading to the neglect of general oral health. This avoidance is often amplified by the fear of potential pain and dissatisfaction after a dental appointment. A music listening intervention could be beneficial to reduce anxiety, pain and dissatisfaction. This intervention has the advantage to be non-invasive, cheap, and easy to implement in clinical settings. The objective of this study is to explore the effects of a personalised musical intervention on anxiety, pain and dissatisfaction associated with an autogenous gingival graft in comparison to the use of an audiobook (control). In this regard, three groups of patients will receive the gingival graft along with the personalized music intervention (n=20), an audiobook (n=20) or standard care (n=20). Participants will be distributed randomly between conditions in a single blind design (surgeons will be unaware of the condition). However, since the third standard care control group was added as of 07-01-2023, all recruited participants will be enrolled in the standard care control group (non-randomized). Self-reported measures of anxiety, pain, and dissatisfaction will be taken at different times (baseline, preoperative, postoperative, and follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Need a gingival graft that will not exceed 1.5 hour of surgery
* Understand spoken and written French or English
* Has the capacity to understand procedures and follow instructions
* Consent to follow instructions
* Consent to receive either the active or control sound condition
* Being 18 years or older

Exclusion Criteria:

* Do not need a gingival graft
* Need a gingival graft that will last more than 1.5 hour of surgery
* Mental health or neurological disorders
* Auditory disorder
* Allergy or intolerance to NSAIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
burden of care | immediately before surgery
  anxiety, pain and satisfaction measured using VAS scales (0 - 10mm; 0= no anxiety, no pain, no satisfaction, and 10= maximum anxiety, worst pain imaginable, maximum satisfaction)
burden of care | immediately after surgery
  anxiety, pain and satisfaction measured using VAS scales (0 - 10mm; 0= no anxiety, no pain, no satisfaction, and 10= maximum anxiety, worst pain imaginable, maximum satisfaction)
burden of care | 2 weeks postop
  anxiety, pain and satisfaction measured using VAS scales (0 - 10mm; 0= no anxiety, no pain, no satisfaction, and 10= maximum anxiety, worst pain imaginable, maximum satisfaction)

SECONDARY OUTCOMES:
sociodemographic data | 1 week before surgery
  age, sex, gender, level of education, yearly income
participants' expectations | immediately before surgery
  expected pain and complications, expected and felt efficiency of the sound condition (VAS scales) (0 - 10mm; 0= no pain, no complications, no efficiency, and 10= worst pain imaginable, maximum complication, maximum efficiency)
participants' expectations | immediately after surgery
  expected pain and complications, expected and felt efficiency of the sound condition (VAS scales) (0 - 10mm; 0= no pain, no complications, no efficiency, and 10= worst pain imaginable, maximum complication, maximum efficiency)
participants' expectations | 2 weeks postop
  expected pain and complications, expected and felt efficiency of the sound condition (VAS scales) (0 - 10mm; 0= no pain, no complications, no efficiency, and 10= worst pain imaginable, maximum complication, maximum efficiency)
Index of dental anxiety and fear | 1 week before surgery
  A.1. To what extent are you anxious about the following things when you go to the dentist? Not at all A little Somewhat Moderately Very much
  1. Painful or uncomfortable procedures
  2. Feeling embarrassed or ashamed
  3. Not being in control of what is happening
  4. Feeling sick, queasy, or disgusted
  5. Numbness caused by the anesthetic
  6. Not knowing what the dentist is going to do
  7. The cost of dental treatment
  8. Needles or injections
  9. Gagging or choking
  10. Having an unsympathetic or unkind dentist
  A.2 On the following scale, how would you rate your level of anxiety at the present time?
  No anxiety
  Maximum anxiety
  A.3.1 On the following scale, what level of pain do you experience right now? Worst pain
  No pain
  imaginable
  A.3.2 On the following scale, what level of pain do you expect to experience during surgery? Worst pain
  No pain
  imaginable
Index of dental anxiety and fear | immediately before surgery
  A.1. To what extent are you anxious about the following things when you go to the dentist? Not at all A little Somewhat Moderately Very much
  1. Painful or uncomfortable procedures
  2. Feeling embarrassed or ashamed
  3. Not being in control of what is happening
  4. Feeling sick, queasy, or disgusted
  5. Numbness caused by the anesthetic
  6. Not knowing what the dentist is going to do
  7. The cost of dental treatment
  8. Needles or injections
  9. Gagging or choking
  10. Having an unsympathetic or unkind dentist
  A.2 On the following VAS 10-mm scale, how would you rate your level of anxiety at the present time?
  No anxiety
  Maximum anxiety
  A.3.1 On the following VAS 10-mm scale, what level of pain do you experience right now? Worst pain
  No pain
  imaginable
  A.3.2 On the following VAS 10-mm scale, what level of pain do you expect to experience during surgery? Worst pain
  No pain
  imaginable
Index of dental anxiety and fear | immediately after surgery
  A.1. To what extent are you anxious about the following things when you go to the dentist? Not at all A little Somewhat Moderately Very much
  1. Painful or uncomfortable procedures
  2. Feeling embarrassed or ashamed
  3. Not being in control of what is happening
  4. Feeling sick, queasy, or disgusted
  5. Numbness caused by the anesthetic
  6. Not knowing what the dentist is going to do
  7. The cost of dental treatment
  8. Needles or injections
  9. Gagging or choking
  10. Having an unsympathetic or unkind dentist
  A.2 On the following VAS 10-mm scale, how would you rate your level of anxiety at the present time?
  No anxiety
  Maximum anxiety
  A.3.1 On the following VAS 10-mm scale, what level of pain do you experience right now? Worst pain
  No pain
  imaginable
  A.3.2 On the following VAS 10-mm scale, what level of pain do you expect to experience during surgery? Worst pain
  No pain
  imaginable
Index of dental anxiety and fear | 2 weeks postop
  A.1. To what extent are you anxious about the following things when you go to the dentist? Not at all A little Somewhat Moderately Very much
  1. Painful or uncomfortable procedures
  2. Feeling embarrassed or ashamed
  3. Not being in control of what is happening
  4. Feeling sick, queasy, or disgusted
  5. Numbness caused by the anesthetic
  6. Not knowing what the dentist is going to do
  7. The cost of dental treatment
  8. Needles or injections
  9. Gagging or choking
  10. Having an unsympathetic or unkind dentist
  A.2 On the following VAS 10-mm scale, how would you rate your level of anxiety at the present time?
  No anxiety
  Maximum anxiety
  A.3.1 On the following VAS 10-mm scale, what level of pain do you experience right now? Worst pain
  No pain
  imaginable
  A.3.2 On the following VAS 10-mm scale, what level of pain do you expect to experience during surgery? Worst pain
  No pain
  imaginable
State-trait anxiety inventory (Spielberg DC et al, 1977) | 1 week before surgery
  Do not spend too much time on any one statement but give the answer which seems to describe your present feelings best.
  Choice of selection: not at all (1), somewhat (2), moderately so (3), very much (4)
  Right now:
  1. I feel calm
  2. I feel secure
  3. I am tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel comfortable
  11. I feel self-confident
  12. I feel nervous
  13. I am jittery
  14. I feel indecisive,
  15. I am relaxed
  16. I feel content,
  17. I am worried,
  18. I feel confused,
  19. I feel steady
  20. I feel pleasant
State-trait anxiety inventory (Spielberg DC et al, 1977) | immediately before surgery
  Do not spend too much time on any one statement but give the answer which seems to describe your present feelings best.
  Choice of selection: not at all (1), somewhat (2), moderately so (3), very much (4)
  Right now:
  1. I feel calm
  2. I feel secure
  3. I am tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel comfortable
  11. I feel self-confident
  12. I feel nervous
  13. I am jittery
  14. I feel indecisive,
  15. I am relaxed
  16. I feel content,
  17. I am worried,
  18. I feel confused,
  19. I feel steady
  20. I feel pleasant
State-trait anxiety inventory | immediately after surgery
  validated general anxiety questionnaire
State-trait anxiety inventory (Spielberg DC et al, 1977) | 2 weeks postop
  Do not spend too much time on any one statement but give the answer which seems to describe your present feelings best.
  Choice of selection: not at all (1), somewhat (2), moderately so (3), very much (4)
  Right now:
  1. I feel calm
  2. I feel secure
  3. I am tense
  4. I feel strained
  5. I feel at ease
  6. I feel upset
  7. I am presently worrying over possible misfortunes
  8. I feel satisfied
  9. I feel frightened
  10. I feel comfortable
  11. I feel self-confident
  12. I feel nervous
  13. I am jittery
  14. I feel indecisive,
  15. I am relaxed
  16. I feel content,
  17. I am worried,
  18. I feel confused,
  19. I feel steady
  20. I feel pleasant
Anxiety coping strategies | 1 week before surgery
  Q.1: Have you ever used strategies to manage your anxiety at the dentist? __Yes ___No 1. If yes, can you indicate them? ___Do breathing exercises ___Meditate ___Playing sports
  * Talking, writing, or texting to a friend ___Reading ___Listening to music___Watching a movie
  * Playing a game ___Other: ..........................................................................................................................
  Q.2: Did you already have a gingival graft in the past? ___Yes ___No
  1 If yes, in your opinion, how did the intervention go?
  Really bad___ Really good ___
  C2.1.1 Why did you choose this answer? ………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………………
Cafeine and medications consumption | 1 week before surgery
  mean consumption per week, # taken today (coffee, tea, sodas, energy drinks, medications = analgesics, stimulants, nutrition supplements, other medications)
Cafeine and medications consumption | immediately before surgery
  mean consumption per week, # taken today (coffee, tea, sodas, energy drinks, medications = analgesics, stimulants, nutrition supplements, other medications)
Cafeine and medications consumption | 2 weeks postop
  mean consumption per week, # taken today (coffee, tea, sodas, energy drinks, medications = analgesics, stimulants, nutrition supplements, other medications)
Feelings at the present moment | immediately before surgery
  valence, arousal, dominance using numerical and illustrated scales (A to I; A = happy/elated, excited/involved, being controlled/taken care of; I = unhappy/sad, calm/bored, being in control/on top of things)
Feelings at the present moment | immediately after surgery
  valence, arousal, dominance using numerical and illustrated scales (A to I; A = happy/elated, excited/involved, being controlled/taken care of; I = unhappy/sad, calm/bored, being in control/on top of things)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Clinique dentaire Antoine Sabeh, Montreal, Quebec
  - Le Groupe des parodontistes, Montreal, Quebec
  - Université de Montréal - Faculty of Dentistry - Dental clinics, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No